CLINICAL TRIAL: NCT05641662
Title: Heart-eXg Study: Effects of Exergaming to Reduce Sedentary Time in Inactive Patients With Heart Failure: An International Multi-center, Randomized, Parallel-group Study
Brief Title: Effects of Exergaming to Reduce Sedentary Time in Inactive Patients With Heart Failure
Acronym: Heart-eXg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Tiny Jaarsma, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DNR 2020-01109
Record Dates: First submitted 2022-05-17; First posted 2022-12-08 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame group (Experimental): Patients will be introduced to the exergame and the exergame will be installed following a protocol either by the patients themselves or an instructor of the study.
  Patients will be advised to exergame daily based on their activity monitor reading at baseline and based on their current activity level and preferences.
  During the 3 months of active intervention patients will receive feedback on their activity level and data will also be shared with the coach who will use it to adapt the gaming advice. A clear exergaming goal will be set together by patient and coach. In the first month, they will receive weekly feedback on their performance based on the readings from the activity monitor and the reading from the exergame. In the rest of the active study team the frequency of the contact with the coach will be personalized.
  Interventions: Other: Heart Farming
- Control group (No Intervention): Patients will receive a protocol-based activity advice (one time) from the HF team (nurse, cardiologist and/or physiotherapist) that corresponds to the intervention group in terms of time and effort. Participants in the control group are encouraged to decrease their sedentary behaviour to the same extent as the intervention group, and if possible be physical active 30 minutes for 5 days a week.

INTERVENTIONS:
Other: Heart Farming — Heart Farming is a mobile game. which can be played indoors and outdoors and stimulates players to be physically active. The game is built around a theme (farming) and users are challenged to collect products by being active. The phone will register movements and convert them into points and fruits and vegetables. For the basic playing only 10 minutes walking a day with the game is possible and is rewarded. For players who want more challenge and level of trading products and collecting products in groups is added. The game is adaptable to different levels of mobility and players can invite others to play with them. Players can see their own game results, progression, and active time.
  Arms: Exergame group

SUMMARY:
The goal of this to determine the effect of tailored exergaming for inactive patients with heart failure to reduce their sedentary time, improve their daily physical activity, exercise capacity, decrease frailty and improve health-related quality of life.

Participants will, on a background of standard guideline-directed medical therapy patients, be randomised to tailored activity advice (control) or the Heart-Exergame (Heart-eXg) intervention for a period of 3 months. Patients randomised to the Heart-eXg group will receive an exergame with feedback and tailoring to adapt the exergaming advice. Patients will also be able to play with a person in their own network.

DETAILED DESCRIPTION:
Rationale: Heart failure (HF) is an increasing global health concern with over 20 million patients worldwide. A decrease in sedentary time can have beneficial effects for a growing group of inactive patients with HF. The use of exergames (games to improve physical activity) is promising for people who are home bound and physically inactive. Such a gaming activity should be attractive, tailored to preferences and to capacity.

Objective: To determine the effect of tailored exergaming for inactive patients with HF to reduce their sedentary time, improve their daily physical activity, exercise capacity, decrease frailty and improve health-related quality of life.

Study design: A pilot study and a multicentre, open-label 1:1 randomised clinical trial with 6 months follow-up.

Study population: Adult patients with symptomatic HF: n= 20 for the pilot study and n=600 for the main study

Intervention: On a background of standard guideline-directed medical therapy patients will be randomised to tailored activity advice (control) or the Heart-Exergame (Heart-eXg) intervention for a period of 3 months. Patients randomised to the Heart-eXg group will receive an exergame with feedback and tailoring to adapt the exergaming advice. Patients will also be able to play with a person in their own network.

Main study parameters/endpoints: Primary endpoint is sedentary time (actigraphy). Secondary outcomes are daily physical activity, submaximal exercise capacity, physical frailty, health-related quality of life.

This study will gain insight into the effects of using an exergame that is easily applicable and affordable. Given the vast growing target population of patients with HF worldwide, and the simplicity of the intervention, potentially millions of patients may benefit from the results of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with symptomatic HF (NYHA II-IV) as diagnosed by cardiologist, (independent of Ejection Fraction: Patients with a preserved ejection fraction (HFpEF), mid-range ejection fraction (HFmrREF) or reduced ejection fraction (HFrEF) can be included.
2. Clinically stable
3. Physically inactive
4. Older than 18 years, there is no upper age limit,
5. Speak/understand the language of the country where the study is taking place.
6. Wanting to use a smartphone for the study (if patients do not have a smartphone, they can borrow it from the study team for the duration of the study)

Exclusion Criteria:

1. Unable to use an exergame due to visual, hearing, cognitive impairment assessed by HF nurse or cardiologist.
2. Not being able to perform the 6-minute walk test.
3. Not being able or willing to wear an activity monitor.
4. Currently included in a rehabilitation program
5. Lack of willingness to play an exergame.
6. Co-morbidity that hinders benefitting for this form of exercise (history of stroke, severe cognitive dysfunction, or a life expectancy shorter than 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-08-16 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Sedentary time | 3 months
  Sedentary time measured with activity monitor Actigraph

SECONDARY OUTCOMES:
Exercise Capacity | Baseline, 3 months and 6 months
  6-minute walk test
Frailty | Baseline, 3 months and 6 months
  Fried Frailty tests
Clinical frailty | Baseline, 3 months and 6 months
  Clinical Frailty Scale: a frailty score ranging from 1 (very fit) to 9 (terminally ill)
Heart Failure specific Quality of Life | Baseline, 3 months and 6 months
  12 item Kansas City Cardiomyopathy includes that quantifies physical limitations, symptom frequency, Quality of Life, and social limitation, along with a summary scores for each domain, scoring from 0 to 100. Zero denoting the worst and 100 the best possible health status.
General Quality of Life | Baseline, 3 months and 6 months
  EuroQol-5 Dimension 5 levels (EQ-5D) includes five domain scales (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and five levels for each domain. A higher score in the EQ-5D-5L indicated better HRQOL
Sedentary time | 6 months
  Sedentary time measured with activity monitor Actigraph

OTHER OUTCOMES:
Patient expectations | Baseline and 6 months
  Open ended interview questions
Exercise motivation | Baseline, 3 months and 6 months
  The situational motivation scale (SIMS): 16 items measuring four forms of motivation with exh four items (amotivation, external, identified, and intrinsic motivation). Each item is rated on a 7-point Likert scale ranging from 1 "corresponds not at all" to 7 "corresponds exactly." The score of each form of motivation ranges from 4-28, with a higher score meaning higher motivation.
Cost | 6 months
  Cost logbook
Willingness to pay | 6 months
  Interviews
Time exergaming | During the 6 months intervention
  Record time exergaming
Enjoyment physical activity | 3 and 6 months in the intervention group only
  Exergaming Enjoyment Scale, 20 items, scoring ranging from 20-100
Cognitive function | Baseline, 3 months and 6 months
  Montreal Cognitive Assessment (MoCA)
Social and daily function | Baseline, 3 months and 6 months
  Canadian Occupational Performance Measure (COPM)
Depression | Baseline, 3 months and 6 months
  Hospital Anxiety and Depression scale( HADs): two conjoint 7-item subscales, one specifically targeted at anxiety (HADS-A) and one focussing on depression (HADS-D). Raw scores of between 8 and 10 identify mild cases of depression or anxiety, 11-15 moderate cases, and 16 or above, severe cases.
Self-care | Baseline, 3 months and 6 months
  European Self-Care Behavioural Scale (ESCBS): nine statements about HF-specific self-care which have to be rated on a 5-point Likert scale ('completely agree' and 'I don't agree at all').The sum score of range from 9 to 45, with lower scores indicating better self-care.
Knowledge | Baseline
  Heart Failure Knowledge Scale: 15-item, self-administered questionnaire that covers items concerning HF knowledge in general, knowledge on HF treatment (including diet and fluid restriction) and HF symptoms and symptom recognition. The scale has a minimum score of 0 (no knowledge) and a maximum score of 15 points (optimal knowledge).
Clinical Data | Baseline
  Clinical data from patient journal
Adverse events | Throughout the trial of 6 months
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tiny Jaarsma, PhD, Principal Investigator — Linkoeping University
Locations (10):
- P. J. Safarik University, Norrköping, Slovakia
- Spain (5):
  - Germans Trias i Pujol Hospital, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital del Mar, Barcelona
  - Xarxa Assistencial Universitaria, Manresa
  - INCLIVA, Valencia
- Sweden (4):
  - Jönköping Hospital Rydhov, Jönköping
  - Kalmar Länssjukhuset, Kalmar
  - Linköping University Hospital, Linköping
  - Primary Health Care Centers Östergötland, Norrköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — http://www.heart-exg.com/index.php